CLINICAL TRIAL: NCT00102752
Title: A Phase 1/2 Dose-Escalation Study of the Safety, Efficacy and Pharmacokinetics of Glufosfamide in Combination With Gemcitabine in Advanced Solid Tumors and Pancreatic Adenocarcinoma
Brief Title: Study of Safety and Efficacy of Glufosfamide in Combination With Gemcitabine in Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Threshold Pharmaceuticals (Industry)
Collaborators: PPD Development, LP (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH-CR-301
Record Dates: First submitted 2005-02-01; First posted 2005-02-02 (Estimated); Last update posted 2009-04-30 (Estimated); Status verified 2009-04

CONDITIONS: Neoplasms; Pancreatic Neoplasms
Keywords: Pancreas; Cancer; Metastatic; Glufosfamide; Advanced; Solid; Tumor; Advanced Solid Tumors; Pancreatic Adenocarcinoma
MeSH Terms: conditions — Neoplasms; Pancreatic Neoplasms; Neoplasm Metastasis | interventions — beta-D-glucosylisophosphoramide mustard; Gemcitabine

INTERVENTIONS:
Drug: Glufosfamide
Drug: Gemcitabine

SUMMARY:
The purpose of this study is to determine the safety of glufosfamide when administered in combination with gemcitabine.

DETAILED DESCRIPTION:
This study, TH-CR-301, is a Phase 1/2 study that will evaluate the efficacy and safety of glufosfamide in combination with gemcitabine in advanced solid tumors or in first line treatment of pancreatic cancer.

Study Hypothesis: Glufosfamide in combination with gemcitabine may provide benefits in survival to patients with advanced solid tumors or metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Histologically or cytologically confirmed, locally advanced or metastatic solid malignancy; previously treated with at least one chemotherapy regimen for advanced or metastatic disease or no effective standard treatment is available OR
* Metastatic and/or locally advanced, inoperable pancreatic adenocarcinoma proven either by histology (surgical biopsy) or cytology (CT- or endoscopic-guided)
* Measurable or nonmeasurable disease by RECIST criteria (at least one target or nontarget lesion)
* Recovered from reversible toxicities of prior therapy
* Karnofsky performance status ≥70
* Women of childbearing potential and men to use effective means of contraception from entry into the study through 6 months after the last dose
* Ability to understand the purposes and risks of the study and provide written informed consent.

Exclusion Criteria:

* Prior chemotherapy for metastatic/locally advanced pancreatic cancer
* Prior administration of gemcitabine
* Radiation therapy within 28 days prior to study start
* Hormonal therapy, biologic therapy, chemotherapy or other systemic anti-tumor therapy for cancer within 21 days prior to study start
* Symptomatic brain metastases (baseline CT scan is not required in asymptomatic subjects)
* Active, clinically significant infection requiring antibiotics
* Known HIV positive or active hepatitis B or C
* History or symptoms of cardiovascular disease (NYHA Class 3 or 4)
* Other primary malignancies (other than treated non-melanoma skin cancer or treated in situ cancer) within the past 5 years
* Major surgery within 3 weeks of the start of study treatment, without complete recovery
* Clinically significant abnormalities in laboratory test results (including complete blood count, chemistry panel including electrolytes, and urinalysis)

  * Hemoglobin <9 g/dL (may receive transfusion or erythropoietin to maintain),
  * ANC <1500/μL,
  * Platelet count <100,000/μL,
  * Total bilirubin > 1.5 ×ULN,
  * AST/ALT > 2.5-fold above ULN (>5-fold above ULN if liver metastases),
  * Serum creatinine > 2 mg/dL,
  * Creatinine clearance < 60 mL/min (calculated)
* Females who are pregnant or breast-feeding
* Participation in an investigational drug or device study within 28 days of the first day of dosing on this study
* Concomitant disease or condition that could interfere with the conduct of the study
* Unwillingness or inability to comply with the study protocol for any other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47
Dates: Start 2004-12; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Overall objective response rate

SECONDARY OUTCOMES:
Overall survival
6- and 12- month survival
Progression-free survival
Duration of objective response
Serum CA-19-9

CONTACTS AND LOCATIONS:
Locations (9):
- United States (3):
  - Arizona Cancer Center, Tucson, Arizona
  - Indiana Cancer Center, Indianapolis, Indiana
  - Norton Healthcare Cancer Center, Louisville, Kentucky
- Brazil (6):
  - Hospital de Doenças Cardiovasculares - Biocor, Nova Lima, BH
  - Hospital Mãe de Deus, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceição, Porto Alegre, Rio Grande do Sul
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos, São Paulo
  - Universidade Federal de São Paulo - Hospital São Paulo, São Paulo, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo, São Paulo

REFERENCES:
- See also: Threshold Pharmaceuticals Website — http://www.thresholdpharm.com